CLINICAL TRIAL: NCT07372404
Title: The Effect of Allogeneic Human Fat-Derived Extract on Skin Graft Donor Site Wound Healing
Brief Title: Allogeneic Adipose Tissue Extract in Wound Treatment and Scar Maturation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linio Biotech Oy (Industry)
Collaborators: Hospital Nova of Central Finland (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-003
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-10

CONDITIONS: Wound Healing
Keywords: allogeneic tissue product; adipose-derived tissue; skin graft donor site; split-thickness skin graft; epithelialization; wound assessment; scar quality; scar maturation; scar thickness
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants are not randomized into different arms. Each participant will have two skin graft donor sites harvested. One donor site wound will be treated topically with adipose tissue extract immediately after harvesting and again on Day 3, while the other donor site wound will receive standard care. Photographic documentation and clinical evaluation of the donor site wounds will be performed on Days 3, 7, 14, and 60 to monitor wound healing progression. Study participants and independent evaluators are blinded to treatment allocation.
Masking Description: Participants and outcome independent evaluators are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adipose tissue extract treatment (Experimental): Study participants will have two skin graft donor sites harvested. One donor site will be treated topically with adipose tissue extract immediately after harvesting and again on Day 3. The other skin graft donor site wound will receive standard of care, following the hospital's Current Care Guidelines.
  Interventions: Procedure: Topical treatment

INTERVENTIONS:
Procedure: Topical treatment — The adipose tissue extract will be applied topically to one skin graft donor site wound immediately after harvesting and reapplied on Day 3. The other donor site will receives standard wound care according to hospital protocol, without application of adipose tissue extract. Wounds will be photographed and assessed on Days 3, 7, 14, and 60. Study participants and independent evaluators are blinded to treatment allocation.

SUMMARY:
This study will evaluate the effect of an allogeneic adipose tissue extract on wound healing and scar maturation. Thirty adult patients scheduled for skin graft surgery will be enrolled. Each patient will have two skin graft donor sites harvested. One skin graft donor site wound will be treated topically with the adipose tissue extract, applied immediately after harvesting and reapplied on Day 3, while the other skin graft donor site wound will receive standard care. The main outcome is the time to complete epithelialization of the wound, as confirmed by investigators and independent reviewers. Secondary measures include wound characteristics, scar formation and scar quality, and monitoring of adverse events, such as wound deterioration.

DETAILED DESCRIPTION:
Cell-free preparate of human adipose tissue is intended to be used in the human body for its original purpose to supplement and replace local extracellular matrix deficiencies in soft tissue, including skin. The tissue product provides a temporary conductive environment into the injured area. This facilitates the ability of local cells to re-populate the damaged soft tissue and skin area, thereby enabling the deposition of extracellular matrix and repair of the tissue.

ELIGIBILITY:
Inclusion Criteria:

* Wound of at least 10 cm3 with an indication of skin graft surgery (two skin grafts harvested and used)
* Adult (age 18 years or more)
* Able and willing to give informed consent
* Reasonably accessible to the study clinic and compliant to wound treatment

Exclusion Criteria:

* Known allergy to any of the preparation used in the study (Tience)
* Systemic cancer (does not include carcinoma in situ of the cervix or local skin cancers such as basiloma)
* Pregnancy or nursing
* Those who withhold consent
* Active infection on the receptor site, donor site or sepsis
* Any other serious disease likely to compromise the outcome of the trial, such as critical renal disease (creatinine greater than 300 mmol/l)
* Those living at such a distance from the clinic as would make frequent assessment visits inappropriately expensive and/or impractical.
* Those with conditions, which tend to limit a patient´s ability or willingness to restrict activities or comply with the instructions during the treatment and follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation | Day 3, Day 7, Day 14, Day 60
  The primary efficacy end point will the wound healing time during this study period, in days. Healing will be defined as complete epithelialization (mm paper, photographs), confirmed by an investigator and independent evaluators. The comparison will be made between the donor site treated with allogeneic adipose tissue extract (ATE) and the untreated donor site (standard care) within the same participant.
The number adverse events, including deterioration of the wounds during the study. | Day 3, Day 7, Day 14, Day 60
  The primary safety end points will be the number adverse events, including deterioration of the wounds during the study.
  * Adverse events, including deterioration of wounds
  * Severe wound complications (necrosis, infection)
Clinical evaluation | Day 3, Day 7, Day 14
  The donor site wound physical characteristics will be recorded: moisture, colour, infection and hypergranulation
Clinical imaging | Post op, Day 3, Day 7, Day 14, and Day 60
  Digital photographs will be taken to document the progression of wound healing. One or two blinded plastic surgeons, with no conflicts of interest, will evaluate the donor site wounds and scars based on these photographs. They will assess and compare the donor sites treated with allogeneic adipose tissue extract (ATE) and those treated with standard care, as well as the resulting scars, using the photographic documentation.
Clinical evaluation | Day 60
  Scar scaling, modified Vancouver burn scale consists of six items. All items are scored on a scale ranging from 1 ('like normal skin') to 3 ('worst scar imaginable'). • Vascularity category: pale, pink, red, normal • Pigmentation category: hypo, hyper, normal • Height: plane, depressed, elevated • Matte vs. shine: shine, matte • Contour: forms part of the adjacent skin, small indentation or invagination • Texture: normal, barely palpable, rough, indented

SECONDARY OUTCOMES:
Pain Intensity Measure | Day 3, Day 7, Day 14
  VAS Visual analogue scale (0-10 points)
Clinical evaluation | Day 60
  Scar quality will be assessed using the Patient and Observer Scar Assessment Scale (POSAS), a validated tool that evaluates scars from both the clinician's and the patient's perspectives. The POSAS scale includes seven parameters-each rated from 1 (normal skin) to 10 (worst scar imaginable). The Scale assesses pain, itching, color, stiffness, thickness, irregularity, and overall impression.
Fever (only symptomatic patients) | Day 3, Day 7, and Day 14
  Temperature (°C)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nova, Jyväskylä, Finland, Finland

IPD SHARING:
Plan to Share IPD: Undecided